CLINICAL TRIAL: NCT05553457
Title: MyHand-SCI: a Wearable Robotic Hand Orthosis for C6-C7 Spinal Cord Injury
Brief Title: MyHand-SCI: an Active Hand Orthosis for Spinal Cord Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Joel Stein, MD, Professor and Chair of the Department of Rehabilitation and Regenerative Medicine, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AAAU2339; R01NS115652 (NIH)
Record Dates: First submitted 2022-09-21; First posted 2022-09-23 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Spinal Cord Injuries; Tetraplegia
Keywords: Spinal Cord Injuries; Tetraplegia; Rehabilitation; Robotics; Assistive Technology; Wearable Devices
MeSH Terms: conditions — Spinal Cord Injuries; Quadriplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- MyHand-SCI Device Testing (Experimental): Subjects will attend 1-20 sessions (of approximately 90 mins) to trial a variety of the MyHand-SCI device controls and/or components. Participants will practice various grasp and release activities with the device
  Interventions: Device: Testing of MyHand-SCI Device

INTERVENTIONS:
Device: Testing of MyHand-SCI Device — Subjects will attend 1-20 sessions (approximately 90 minutes) to trial the MyHand-SCI device, including a variety of controls and components.

SUMMARY:
The purpose of this study is to develop and test the hardware and software components of the MyHand-SCI device to assist with hand function for individuals with C6-C7 spinal cord injury.

DETAILED DESCRIPTION:
The purpose of this study is to develop and test the hardware and software components of the MyHand-SCI device to assist with hand function for individuals with C6-C7 spinal cord injury. This is a non-randomized exploratory study to determine feasibility of device use, provide user feedback on device features and function to allow further refinement of the device, and assess the utility and responsiveness of several clinical outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with C6-C7 spinal cord injury, at least 6-months post-injury with impaired upper limb function
* Substantially reduced motor control and strength below the level of their SCI with regard to hand and finger function
* Able to provide informed consent

Exclusion Criteria:

* Fixed upper limb contractures that limit functional use of the hand and arm or ability to use the device
* Severe spasticity (modified Ashworth >2) at elbow, wrist, or fingers
* Any open wounds or unusual skin fragility
* Persistent severe pain in their upper limb

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-10-04 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
System Usability Scale | Up to 2 years at study completion
  The System Usability Scale (SUS) is a reliable tool for measuring the usability of products, including medical devices. It consists of a 10 item questionnaire with five response options (Strongly agree to Strongly disagree).

CONTACTS AND LOCATIONS:
Overall Officials: Joel Stein, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No